CLINICAL TRIAL: NCT02120937
Title: Neural Basis of Mindfulness in Mood Dysregulated Youth
Brief Title: Mindfulness in Mood Dysregulated Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Melissa Delbello, MD, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0453
Record Dates: First submitted 2014-04-18; First posted 2014-04-23 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2015-09

CONDITIONS: Bipolar Disorder; Mood Disorder; Emotional Disturbance
Keywords: amygdala; mindfulness; mood; emotion; bipolar disorder; parental bipolar disorder; adolescence
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders; Affective Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MBCT-C Therapy (Experimental): Mindfulness Based Cognitive Therapy for Children is a manualized psychotherapeutic intervention that combines mindfulness techniques with certain features of cognitive behavioral therapy. This particular protocol for youth includes weekly group sessions, regular home practice, and the core curriculum of formal mindfulness practices (e.g., body scan, sitting, movement, and walking meditations).
  Interventions: Behavioral: MBCT-C Therapy

INTERVENTIONS:
Behavioral: MBCT-C Therapy — Mindfulness Based Cognitive Therapy for Children is a manualized psychotherapeutic intervention that combines mindfulness techniques with certain features of cognitive behavioral therapy. This particular protocol for youth includes weekly group sessions, regular home practice, and the core curriculum of formal mindfulness practices (e.g., body scan, sitting, movement, and walking meditations).
  Other Names: Mindfulness Based Cognitive Therapy-Children

SUMMARY:
Mindfulness group therapy can help children with mood irregularities and family history of bipolar disorder.

DETAILED DESCRIPTION:
Mindfulness Based Cognitive Therapy (MBCT) is a manualized psychotherapeutic intervention that is a combination of mindfulness techniques and cognitive behavioral therapy. MBCT-C, which is mindfulness based cognitive based therapy for children, involves weekly group sessions, home practice, and the core curriculum of formal mindfulness practices (e.g. body scan, sitting, movement and walking meditations). Group sessions will involve guided meditation practices, instructor-led discussion of experiences and psychoeducation. By fopstering the ability to pay close attention to thoughts, emotions and body sensations, participants learn to make better choices to deal with stress, anxiety, depression, pain and other challenges. This can allow them to more effectively use the principles of cognitive behavioral therapy.

Twelve children aged 10-17 with mood dysregulation and a bipolar parent will be in the study for 12 weeks. There will be two groups receiving intervention: one group recruited from the community and one group recruited from a known high-risk cohort.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, subjects must meet the following criteria:

1. Ages 10 -17 years; inclusive at the time of consent
2. At least one biological parent with bipolar I disorder, confirmed with the SCID-P/L
3. CDRS-R score > 28 or YMRS score > 12 or ERC score > 36 at screening and baseline since clinically significant elevation on any of these scales suggests mood dysregulation
4. Fluent in English
5. Provision of written informed consent/assent as previously described
6. Agrees to participate in at least 75% of sessions.

Exclusion Criteria:

1. Previously documented diagnosis of mental retardation or an IQ <70
2. Any lifetime DSM-V diagnosis of bipolar disorder, schizophrenia or other psychotic disorder
3. Previous participation in a mindfulness-based treatment, including MBCT-C
4. A substance use disorder (except nicotine or caffeine) within the past 3 months
5. Judged clinically to be at risk from suicide as defined as having active suicidal ideation, intent or plan, or a serious suicide attempt within 30 days, or a baseline CDRS-R suicide score of >3
6. Concurrent treatment with psychotropic medications that have been adjusted during the 30 days prior to screening or are anticipated during the course of study participation
7. Psychotherapy initiated within 2 month prior to screening or plan to initiate psychotherapy during study participation
8. Significant psychiatric symptoms that require hospitalization
9. Mood symptoms resulting from acute medical illness or acute intoxication or withdrawal from drugs or alcohol as determined by medical evaluation or rapid symptom resolution
10. Female patients who are either pregnant or lactating; All girls will have a urine pregnancy test prior to MR scans
11. Any contraindication to an MRI scan (e.g., metal clips, braces or claustrophobia)
12. Neurological disorders (e.g. epilepsy) or severe head trauma resulting in loss of consciousness for > 10 minutes or any unstable medical illness.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2014-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in ERC | 12 weeks
  Change from baseline to endpoint ( 12 weeks) in ratings on the Emotion Regulation Checklist
Change in CDRS-R | 12 weeks
  Change from baseline to endpoint (12 weeks) on the ratings on the Children's Depression Rating Scale-Revised.
Change in YMRS | 12 weeks
  Change from baseline to endpoint (12 weeks) in ratings on the Young Mania Rating Scale.

SECONDARY OUTCOMES:
Change in amygdala, insula, and prefrontal activation. | 12 weeks
  We will examine baseline to endpoint changes in task related VLPFC, amygdala, and insula activation. We will examine associations among changes in activation in these brain regions and changes in mood regulation rating scale scores.Additionally, we will examine changes in seed-based resting state connectivity measures using amygdala and insula as the seeds and examining connectivity with VLPFC regions. Finally, we will use correlation to assess associations among changes in resting state connectivity of these regions and changes in mindfulness measures.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa P DelBello, MD, Principal Investigator — University of Cincinnati; Sian Cotton, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No